CLINICAL TRIAL: NCT01221298
Title: An Open-Label Pilot Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Antiviral Activity of ABT-450 With Ritonavir (ABT-450/r) Dosed in Combination With ABT-072 and Ribavirin (RBV) in Treatment-Naive Subjects With Genotype 1 Chronic Hepatitis C Virus (HCV) Infection
Brief Title: A Pilot Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Antiviral Activity of ABT-450 With Ritonavir (ABT-450/r) Dosed in Combination With ABT-072 and Ribavirin (RBV)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M12-267
Record Dates: First submitted 2010-10-13; First posted 2010-10-15 (Estimated); Results first posted 2015-01-08 (Estimated); Last update posted 2015-01-08 (Estimated); Status verified 2014-12

CONDITIONS: Hepatitis C; HCV; Chronic Hepatitis C Infection; Hepatitis C Genotype 1
MeSH Terms: conditions — Hepatitis C | interventions — paritaprevir; ABT-072; Ribavirin; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ABT-450/r and ABT-072, plus ribavirin (RBV) (Experimental): ABT-450/r (150/100 mg) once daily (QD) and ABT-072 (400 mg) QD plus weight-based RBV divided twice daily (BID) for 12 weeks.
  Interventions: Drug: ABT-450; Drug: ABT-072; Drug: Ribavirin; Drug: Ritonavir

INTERVENTIONS:
Drug: ABT-450 — tablets
Drug: ABT-072 — tablets
Drug: Ribavirin — tablets
Drug: Ritonavir — capsules
  Other Names: Norvir

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics, and antiviral activity of ABT-450 with ritonavir (ABT-450/r) dosed in combination with ABT-072 and ribavirin (RBV) in treatment-naïve participants with genotype 1 chronic hepatitis C virus (HCV) infection.

DETAILED DESCRIPTION:
This was a Phase 2a multicenter, open-label, single arm, combination treatment study of a regimen of ABT-450/r/ABT-072, and ribavirin (RBV) in hepatitis C virus (HCV) genotype 1-(1a or 1b) infected treatment-naïve participants.

ELIGIBILITY:
Inclusion Criteria:

* Chronic hepatitis C, genotype 1 infection with interleukin 28B (IL28B) rs12979860 genotype C/C.
* Liver biopsy within 3 years with histology consistent with hepatitis C virus (HCV) - induced liver damage, with no evidence of cirrhosis or liver pathology due to any cause other than chronic HCV.
* Treatment naïve male or female between the ages of 18 and 65.
* Females must be postmenopausal for at least 2 years or surgically sterile.
* Be in a condition of general good health, as perceived by the investigator, other than hepatitis C virus infection.
* Body mass index 18 to < 35 kg/m^2 .

Exclusion Criteria:

* Significant sensitivity to any drug.
* Use of herbal supplements within 2 weeks prior to study drug dosing.
* Positive screen for certain drugs or alcohol.
* Positive hepatitis B surface antigen or anti-human immunodeficiency virus (HIV) antibody.
* Use of strong cytochrome P450 3A (CYP3A), cytochrome P450 2C8 (CYP2C8), and organic anion transporting polypeptide 1B1 (OATP1B1) enzyme inducers or inhibitors within 1 month of dosing.
* Prior treatment with any investigational or commercially available anti-hepatitis C virus agents.
* Abnormal laboratory tests.
* Cirrhosis or extensive bridging fibrosis.
* History of cardiac disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2010-10; Primary Completion 2011-05 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Cohen, MD, Study Director — AbbVie
Locations (4):
- United States (4):
  - Site Reference ID/Investigator# 41128, Los Angeles, California
  - Site Reference ID/Investigator# 42262, Chicago, Illinois
  - Site Reference ID/Investigator# 41127, San Antonio, Texas
  - Site Reference ID/Investigator# 43182, Seattle, Washington

REFERENCES:
- [Derived] Lawitz E, Poordad F, Kowdley KV, Cohen DE, Podsadecki T, Siggelkow S, Larsen L, Menon R, Koev G, Tripathi R, Pilot-Matias T, Bernstein B. A phase 2a trial of 12-week interferon-free therapy with two direct-acting antivirals (ABT-450/r, ABT-072) and ribavirin in IL28B C/C patients with chronic hepatitis C genotype 1. J Hepatol. 2013 Jul;59(1):18-23. doi: 10.1016/j.jhep.2013.02.009. Epub 2013 Feb 22. PMID 23439262
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ABT-450/r and ABT-072, Plus Ribavirin (RBV)
Started | 11
Completed | 11 (The number of participants who completed study drug)
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Baseline analyses included all participants.
Arm/Group | ABT-450/r and ABT-072, Plus Ribavirin (RBV)
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.4 (7.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 8
Hepatitis C Virus (HCV) Genotype/ Subtype [Number; unit: participants]
  1A | 8
  1B | 3
Interleukin 28B (IL28B) Genotype [Number; unit: participants]
  CC | 11
  CT | 0
  TT | 0
  Missing | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) Suppressed Below the Lower Limit of Quantitation (LLOQ) From Week 4 Through Week 12
Description: Analysis of the percentage of participants with hepatitis C virus ribonucleic acid less than the lower limit of quantitation (< 25 IU/mL).
Time Frame: Week 4 through Week 12
Population: For the percentage of subjects with HCV RNA suppressed below the LLOQ from Week 4 through Week 12 out of all subjects dosed, it was assumed that if 60% of subjects were successfully suppressed from Week 4 through Week 12 then 20 subjects would give a 95% two-sided confidence interval of (36.1%, 80.9%) using binomial exact methods.
Measure: Number; unit: percentage of participants
Arm/Group | ABT-450/r and ABT-072, Plus Ribavirin (RBV)
Number analyzed (Participants) | 11
percentage of participants | 100

2. Secondary Outcome: Percentage of Participants With Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) < 1000 International Units Per Milliliter (IU/mL)
Description: Analysis of participants with HCV RNA levels below 1000 IU/mL at Week 2.
Time Frame: Week 2
Population: Efficacy analyses included all participants who received at least 1 dose of study drug (ITT). Participants with missing data were imputed as failures.
Measure: Number; unit: percentage of participants
Arm/Group | ABT-450/r and ABT-072, Plus Ribavirin (RBV)
Number analyzed (Participants) | 11
percentage of participants | 100

3. Secondary Outcome: Percentage of Participants With Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) Below the Lower Limit of Quantitation (LLOQ) at Week 4
Description: Analysis of percentage of participants with hepatitis C virus ribonucleic acid less than the lower limit of quantitation (< 25 IU/mL).
Time Frame: Week 4
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | ABT-450/r and ABT-072, Plus Ribavirin (RBV)
Number analyzed (Participants) | 11
percentage of participants | 100

4. Secondary Outcome: Percentage of Participants With Sustained Virologic Response 12 Weeks (SVR12) Post-treatment
Description: Sustained Virologic Response 12 (SVR12) is defined as plasma hepatitis C virus ribonucleic acid (HCV RNA) less than the lower limit of quantification (< LLOQ; < 25 IU/mL) 12 weeks after the last dose of study drug.
Time Frame: Post-treatment Day 1 to Post-treatment Week 12
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | ABT-450/r and ABT-072, Plus Ribavirin (RBV)
Number analyzed (Participants) | 11
percentage of participants | 90.9

5. Secondary Outcome: Percentage of Participants With Sustained Virologic Response 24 Weeks (SVR24) Post-Treatment
Description: Sustained Virologic Response 24 (SVR24) is defined as plasma hepatitis C virus ribonucleic acid (HCV RNA) less than the lower limit of quantification (LLOQ; < 25 IU/mL) 24 weeks after the last dose of study drug.
Time Frame: Post-treatment Day 1 to Post-treatment Week 24
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | ABT-450/r and ABT-072, Plus Ribavirin (RBV)
Number analyzed (Participants) | 11
percentage of participants | 90.9

6. Secondary Outcome: Time to Failure to Suppress or Rebound During Treatment
Description: The time to failure to suppress was defined as first day a participant met any virologic stopping criteria during treatment. The virologic stopping criteria also includes failure to achieve a 2 log10 IU/mL decrease in HCV RNA by Week 1, failure to achieve HCV RNA <LLOQ by Week 6, or rebound, defined as first day of 2 consecutive increases of at least 0.5 log10 IU/mL above nadir (local minimum value) or confirmed HCV RNA > lower limit of detection (LLOD) for participants who previously achieved HCV RNA < LLOD.
Time Frame: Day 1 through Week 12
Population: Efficacy analyses included all participants who received at least 1 dose of study drug (ITT).
Measure: Mean (Standard Error); unit: Days
Arm/Group | ABT-450/r and ABT-072, Plus Ribavirin (RBV)
Number analyzed (Participants) | 11
Days | NA (NA) — The time to failure to suppress or rebound during treatment could not be estimated, as no participant met failure to suppress or rebound criteria.

7. Secondary Outcome: Time to Virologic Relapse Through 24 Weeks Post-treatment
Description: Time to confirmed hepatitis C virus (HCV) ribonucleic acid (RNA) ≥ lower limit of quantitation (LLOQ) (2 consecutive measurements ≥ LLOQ) at any point in the post-treatment period among participants with HCV RNA < LLOQ at the end of treatment.
Time Frame: Post-treatment Day 1 to Post-treatment Week 24
Population: Efficacy analyses included all participants who received at least 1 dose of study drug (ITT) with hepatitis C virus (HCV) ribonucleic acid (RNA) < lower limit of quantitation (LLOQ) at the final treatment visit who completed treatment.
Measure: Mean (95% Confidence Interval); unit: Days
Arm/Group | ABT-450/r and ABT-072, Plus Ribavirin (RBV)
Number analyzed (Participants) | 11
Days | 84 (NA) [NA to NA] — Cannot be estimated as only one participant relapsed.

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from the time of study drug administration to 30 days after last dose of study drug (up to 16 weeks).
Description: Serious Adverse Events were also collected from the time that informed consent was obtained until 30 days after last dose (64 weeks).
Arm/Group | ABT-450/r and ABT-072, Plus Ribavirin (RBV)
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 11/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ABT-450/r and ABT-072, Plus Ribavirin (RBV) (N=11)
VERTIGO (Ear and labyrinth disorders) | 1
VISUAL ACUITY REDUCED (Eye disorders) | 1
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 1
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1
DIARRHOEA (Gastrointestinal disorders) | 1
DYSPEPSIA (Gastrointestinal disorders) | 1
FOOD POISONING (Gastrointestinal disorders) | 1
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 2
NAUSEA (Gastrointestinal disorders) | 3
VOMITING (Gastrointestinal disorders) | 1
FATIGUE (General disorders) | 3
INFLUENZA LIKE ILLNESS (General disorders) | 1
OTITIS MEDIA (Infections and infestations) | 1
POST-TRAUMATIC PAIN (Injury, poisoning and procedural complications) | 1
DIABETES MELLITUS (Metabolism and nutrition disorders) | 1
GOUT (Metabolism and nutrition disorders) | 1
DIZZINESS (Nervous system disorders) | 1
DYSGEUSIA (Nervous system disorders) | 1
HEADACHE (Nervous system disorders) | 4
TENSION HEADACHE (Nervous system disorders) | 1
ANXIETY (Psychiatric disorders) | 1
INSOMNIA (Psychiatric disorders) | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1
DRY SKIN (Skin and subcutaneous tissue disorders) | 3
ECZEMA (Skin and subcutaneous tissue disorders) | 1
PRURITUS GENERALISED (Skin and subcutaneous tissue disorders) | 1
RASH (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.